CLINICAL TRIAL: NCT01889641
Title: Intérêt de l'IL-26 Comme Nouveau Marqueur Biologique du Lupus érythémateux systémique
Brief Title: IL-26 and Systemic Lupus Erythematosus
Status: Terminated | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5504
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Diagnosis of Lupus According to ACR criteriaAgreement for the Blood Sampling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with lupus: Patients with lupus (four levels of activity disease)
- healthy volunteers: Subjects controls

SUMMARY:
Treatment of multisystemic forms of lupus displays severe side effects and limited efficacy, underscoring the need to better dissection of the pathogenic mechanisms. Concordant with preliminary data, IL26 signaling could be impaired in systemic lupus. Moreover, IL 26 could be a marker of the disease activity and then a potential therapeutic target. In the present study, serum IL 26 level in lupus patients and control will be measured.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic of Lupus according to ACR criteria ( four criteria are necessary)
* age > 18 years old

Exclusion Criteria:

* treatment by cyclophosphamide, rituximab, belimumab in the year before inclusion study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Assess serum IL-26 as a biological marker of SLE compared with sera from control subjects | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, Bas Rhin, France